CLINICAL TRIAL: NCT00978458
Title: Phase III Study of Radiation Therapy With or Without Temozolomide for Symptomatic or Progressive Low-Grade Gliomas
Brief Title: Radiation Therapy With or Without Temozolomide in Treating Patients With Low-Grade Glioma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: E3F05; ECOG-E3F05
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Brain and Central Nervous System Tumors; Neurotoxicity
Keywords: neurotoxicity; adult diffuse astrocytoma; adult oligodendroglioma; recurrent adult brain tumor; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neurotoxicity Syndromes; Astrocytoma; Oligodendroglioma; Brain Neoplasms; Glioma | interventions — Temozolomide; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

ARMS (2):
- Arm I (Active Comparator): Patients undergo 3-dimensional conformal or intensity-modulated radiotherapy once daily 5 days a week for 5½ weeks (28 fractions).
  Interventions: Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy
- Arm II (Experimental): Patients undergo radiotherapy as in arm I and receive concurrent oral temozolomide once daily for 5½ weeks. Beginning 28 days after completion of chemoradiotherapy, patients receive oral temozolomide alone once daily on days 1-5. Treatment with temozolomide repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temozolomide; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: temozolomide — Given orally
  Arms: Arm II
Radiation: 3-dimensional conformal radiation therapy — Given once daily 5 days a week for 5½ weeks
Radiation: intensity-modulated radiation therapy — Given once daily 5 days a week for 5½ weeks

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether radiation therapy is more effective when given together with or without temozolomide in treating patients with low-grade glioma.

PURPOSE: This randomized phase III trial is studying radiation therapy so see how well it works when given together with or without temozolomide in treating patients with low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether the addition of temozolomide to fractionated radiotherapy improves the progression-free survival (PFS) of patients with symptomatic or progressive low-grade gliomas.
* To determine whether the addition of temozolomide to fractionated radiotherapy improves the median overall survival (OS) of these patients.

Secondary

* To determine whether combination therapy with temozolomide and radiotherapy improves or maintains cognition and quality of life compared to radiotherapy alone.
* To compare the toxicities (severe or worse [≥ grade 3]) of radiotherapy with vs without temozolomide in these patients.
* To assess the impact of the presence or absence of 1p and 19q deletion on PFS and OS.
* To determine the impact of 1p and 19q status on PFS and OS of patients treated with temozolomide.
* To create a tumor and tissue bank, including plasma and germ line DNA, within the ECOG Pathology Coordinating Office.

OUTLINE: This is a multicenter study. Patients are stratified according to age (< 40 years vs ≥ 40 years), 1p and 19q status (both deleted vs either/both intact vs undeterminable), pre-operative maximum tumor diameter (< 6 cm vs ≥ 6 cm [based on T2 or FLAIR MRI]), Karnofsky performance status (60-70% vs 80-100%), and contrast enhancement on pre-treatment MRI scan (present vs absent). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo 3-dimensional conformal or intensity-modulated radiotherapy once daily 5 days a week for 5½ weeks (28 fractions).
* Arm II: Patients undergo radiotherapy as in arm I and receive concurrent oral temozolomide once daily for 5½ weeks. Beginning 28 days after completion of chemoradiotherapy, patients receive oral temozolomide alone once daily on days 1-5. Treatment with temozolomide repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

Some patients undergo quality-of-life and neurocognitive (e.g., visual scanning speed, divided attention, language, memory, and fine motor skills) assessments at baseline, annually until disease progression, and at the time of disease progression.

Tumor tissue samples are collected at baseline for confirmation of diagnosis and determination of 1p and 19q deletion status. Peripheral blood, serum, and additional tumor tissue samples may be collected for further research studies.

After completion of study treatment, patients are followed up periodically for up to 15 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* supratentorial low-grade glioma, including 1 of the following:

  * Grade 2 astrocytoma
  * Grade 2 oligodendroglioma
  * Grade 2 oligoastrocytoma (mixed glioma containing astrocytoma and oligodendroglioma)
* NOTE: *If the pathology from multiple procedures supports the diagnosis of a brain tumor, the qualifying pathology of grade 2 astrocytoma, oligodendroglioma, or oligoastrocytoma must be the most recent pathological diagnosis; no pathological diagnosis of grade 3 or 4 glioma at any time
* Paraffin-embedded tumor specimen available for submission for confirmation of pathological review and determination of 1p and 19q deletion status
* Patients must currently meet ≥ 1 of the following criteria*:

  * Uncontrolled symptoms, defined as any of the following:

    * Headaches associated with mass effect
    * Uncontrolled seizures despite two different antiepileptic drug regimens (i.e., two antiepileptic drugs tested either sequentially or in combination)
    * Focal neurological symptoms
    * Cognitive symptoms or deficits
  * Tumor progression by serial MRIs, defined as any of the following:

    * New or progressive enhancement
    * New or progressive T2 or FLAIR signal abnormality
  * Age ≥ 40 years
* NOTE: *Patients < 40 years of age whose only symptom of low-grade glioma is seizures that are well-controlled on antiepileptic drugs AND who have no evidence of radiographic progression are not eligible.
* Patients who have undergone gross total resection and have no detectable residual disease are eligible
* No pilocytic astrocytoma, ganglioglioma, pleomorphic xanthoastrocytoma, or dysembryoplastic neuroepithelial tumors

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* WBC ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hematocrit ≥ 30%
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Creatinine ≤ 2.0 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Able to undergo MRI with and without contrast
* No other malignancy within the past 5 years, except for nonmelanoma skin cancer or cervical carcinoma in situ
* No uncontrolled infection
* No known HIV positivity
* No medical disorder that would increase risks associated with radiotherapy and temozolomide
* No other disorder that would limit life expectancy to < 5 years

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy, cytotoxic chemotherapy, radiosurgery, or investigational therapy directed at the brain tumor

  * Any number of prior surgical procedures for the brain tumor allowed
* No prior radiotherapy to the head unless the radiotherapy ports entirely excluded the brain
* At least 2 weeks since any prior brain surgery (e.g., stereotatic biopsy, open biopsy, or resection)
* At least 6 weeks since prior MRI and chest x-ray

  * If resection is performed, an MRI after surgery is required

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2009-11-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS)
Overall survival (OS)

SECONDARY OUTCOMES:
Quality of life as assessed by the FACT-BR questionnaire at baseline, annually until disease progression, and at the time of disease progression
Neurocognitive functioning as assessed at baseline, annually until disease progression, and at the time of disease progression
Correlation of pre-treatment 1p and 19q levels in tumor tissue samples with PFS and OS

CONTACTS AND LOCATIONS:
Overall Officials: David Schiff, MD, Study Chair — University of Virginia
Locations (168):
- United States (168):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Community Regional Cancer Care at Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital North, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Norton Suburban Hospital, Louisville, Kentucky
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Billings Clinic - Downtown, Billings, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Oncology Hematology, PC at Albany Medical Center, Albany, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Greer Radiation Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin